CLINICAL TRIAL: NCT02169284
Title: Phase II Clinical Chemoprevention Trial of Weekly Erlotinib Before Bladder Cancer Surgery
Brief Title: Erlotinib Hydrochloride in Treating Patients With Bladder Cancer Undergoing Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2014-01320; NCI-2014-01320 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HHSN261201200033I; N01-CN-2012-00033; CO12336 (Other: University of Wisconsin Hospital and Clinics); UWI2013-01-02 (Other: DCP); N01CN00033 (NIH); P30CA014520 (NIH)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Bladder Carcinoma; Recurrent Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (erlotinib hydrochloride) (Experimental): Patients receive erlotinib hydrochloride PO QD on days 1, 8, and 15. Patients then undergo TURBT or cystectomy on day 16.
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery
- Group II (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1, 8, and 15. Patients then undergo TURBT or cystectomy on day 16.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
  Arms: Group I (erlotinib hydrochloride)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Therapeutic Conventional Surgery — Undergo TURBT or cystectomy

SUMMARY:
This randomized phase II trial studies how well erlotinib hydrochloride works in treating patients with bladder cancer undergoing surgery. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if there is a difference in EGFR phosphorylation in normal appearing bladder epithelium adjacent to tumor approximately 9-18 hours post-study dose, between patients randomized to erlotinib hydrochloride (erlotinib) weekly as compared to placebo.

SECONDARY OBJECTIVES:

I. Assess the tolerance of high dose weekly erlotinib compared to placebo. II. Assess the expression of phosphorylated EGF receptor in tumor tissue when available.

III. Assess the expression of e-cadherin and Ki67 in normal and abnormal urothelium.

IV. Assess the expression of phosphorylated ERK in normal and abnormal urothelium.

V. Assess limited pharmacokinetics of weekly erlotinib. VI. Assess the expression of p53 in normal and abnormal urothelium. VII. Assess the expression of let-7 in normal and abnormal urothelium. VIII. Exploratory assessment of urination symptoms in men.

OUTLINE: Patients are randomized to 1 of 2 treatment groups.

GROUP I: Patients receive erlotinib hydrochloride orally (PO) once daily (QD) on days 1, 8, and 15. Patients then undergo transurethral resection of bladder tumor (TURBT) or cystectomy on day 16.

GROUP II: Patients receive placebo PO QD on days 1, 8, and 15. Patients then undergo TURBT or cystectomy on day 16.

After completion of study treatment, patients are followed up for 7-14 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed or suspected invasive or non-invasive bladder tumor (initial or recurrent) discovered on cystoscopy or radiologic imaging performed within 120 days of randomization
* Patients with muscle invasive bladder cancer (MIBC) must have never received and currently be ineligible for cisplatin-based neoadjuvant chemotherapy due to any of the following:

  * Calculated creatinine clearance of < 60 ml/min
  * Karnofsky performance status (KPS) < 80
  * Solitary kidney or
  * Patient refusal to undergo neoadjuvant chemotherapy
* The participant may have prior treatment for bladder tumor (excluding radiation therapy) provided that treatment:

  * Was completed greater than 30 days prior to the first dose of study agent
* Participants must be a candidate for a trans-urethral resection of the bladder tumor (TURBT), cystectomy (partial or radical) or cystoscopy with biopsy at a participating organization
* Karnofsky >= 60%
* White blood cells (WBC) >= 3000/mm^3
* Platelets >= 100,000mm^3
* Hemoglobin > 10 g/dL
* Alkaline phosphatase =< 1.5 x upper limit of normal
* Bilirubin =< 1.5 x upper limit of normal
* Aspartate aminotransferase (AST) =< 1.5 x upper limit of normal
* Alanine aminotransferase (ALT) =< 1.5 x upper limit of normal
* Bilirubin for Gilbert's =< 3.0 mg/dl
* A calculated creatinine clearance (Cockcroft Gault) of >= 30 ml/min
* Sodium >= 130 mg/dl and =< upper limit of normal
* Potassium >= 3.0 mg/dl and =< upper limit of normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any treatment for the bladder tumor other than intravesical therapy between the pre-study cystoscopy or radiologic imaging which identified the suspected bladder tumor and the scheduled surgical removal or cystoscopy-guided biopsy of that tumor
* Any chemotherapy and/or radiation therapy received =< 3 months of study entry and any immunotherapy received =< 6 months of study entry (with the exception of Bacillus Calmette-Guerin [BCG] treatment)
* Any prior external beam radiation to the pelvis
* A concurrent skin rash or skin condition requiring treatment with a prescription medication
* The following medications may not be taken within 24 hours of the first dose of study agent or at any time while a participant is taking study agent

  * Coumadin
  * Strong CYP3A4 inhibitors including ketoconazole, atazanavir, boceprevir, ceritinib, clarithromycin, cobicistat, darunavir, dasabuvir, idelalisib, indinavir, itraconazole, lopinavir, nefazodone, nelfinavir, ombitasvir, paritaprevir, posaconazole, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole, and grapefruit or grapefruit juice
  * CYP3A4 inducers including rifampicin, rifabutin, rifapentine, phenytoin, carbamazepine, phenobarbital, primidone, enzalutamide, fosphenytoin, lumacaftor, mitotane, and St. John's wort
  * Agents which decrease gastric acid are allowed but should be avoided if possible
  * Participants may resume inhibitors or inducers of CYP3A4 > 14 days after their last dose of study agent
* Participants requiring daily use of non-steroidal anti-inflammatory drugs (NSAIDs), with the exception of =< 81 mg aspirin per day; during study participation, acetaminophen is preferred for treatment of pain; the use of NSAIDs, as needed for pain, is discouraged
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib or clindamycin (topical agent for potential skin toxicity)
* An underlying predisposition to rectal or gastrointestinal bleeding or uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Females who are pregnant or lactating may not participate in this study; females of child-bearing potential must have a negative pregnancy test before starting study agent; patients who have had a bilateral oophorectomy, hysterectomy, or are greater than 1 year since their last menses are not considered to be of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Downs, Principal Investigator — University of Wisconsin, Madison
Locations (6):
- United States (6):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Rochester, Rochester, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology San Antonio Research PA, San Antonio, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 were consented, 13 participants ineligible
Groups:
- Group I (Erlotinib Hydrochloride): Participants receive erlotinib hydrochloride PO QD on days 1, 8, and 15. Participants then undergo TURBT or cystectomy on day 16.
- Group II (Placebo): Participants receive placebo PO QD on days 1, 8, and 15. Participants then undergo TURBT or cystectomy on day 16.
Period: Overall Study
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Started | 24 | 13
Completed | 24 | 12
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo) | Total
Number analyzed (Participants) | 24 | 13 | 37
Age, Customized [Mean (Full Range); unit: years]
  Participant Age | 70.25 [51.69 to 86.09] | 69.32 [59.30 to 85.80] | 69.93 [51.69 to 86.09]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 21 | 10 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 23 | 11 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 22 | 13 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 13 | 37
Karnofsky Performance Status [Count of Participants; unit: Participants] — Karnofsky Performance Status classifies participants based on their functional impairment. A score of 80 = Normal activity with effort; some signs or symptoms of disease; 90 = Able to carry on normal activity; minor signs or symptoms of disease; and 100 = Normal no complaints; no evidence of disease.
  Participants
    80 | 1 | 0 | 1
    90 | 4 | 3 | 7
    100 | 19 | 10 | 29
Ever Smoked [Count of Participants; unit: Participants]
  Yes | 21 | 11 | 32
  No | 3 | 2 | 5
Current Smoker [Count of Participants; unit: Participants]
  Yes | 6 | 3 | 9
  No | 18 | 10 | 28
Systolic Blood Pressure [Mean (Full Range); unit: mmHg] | 134.62 [102.00 to 170.00] | 136.69 [105.00 to 171.00] | 135.35 [102.00 to 171.00]
Diastolic Blood Pressure [Mean (Full Range); unit: mmHg] | 76.62 [57.00 to 94.00] | 78.23 [67.00 to 99.00] | 77.19 [57.00 to 99.00]
Pulse [Mean (Full Range); unit: beats per minute] | 74.75 [56.00 to 101.00] | 69.85 [46.00 to 94.00] | 73.03 [46.00 to 101.00]
Temperature [Mean (Full Range); unit: degrees Fahrenheit] | 97.67 [96.44 to 99.68] | 97.48 [96.00 to 98.42] | 97.61 [96.00 to 99.68]
Height [Mean (Full Range); unit: cm] | 174.77 [152.40 to 187.96] | 174.40 [152.40 to 182.88] | 174.64 [152.40 to 187.96]
Weight [Mean (Full Range); unit: kg] | 89.67 [58.06 to 117.93] | 86.83 [48.99 to 129.27] | 88.67 [48.99 to 129.27]
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 29.37 [22.22 to 48.18] | 28.25 [17.54 to 38.65] | 28.96 [17.54 to 48.18]
Medical History / Baseline Presence of Abnormality or Disease [Number; unit: participants]
  Genitalia | 1 | 2 | 3
  Prostate | 2 | 1 | 3
  Musculoskeletal | 2 | 0 | 2
  Skin | 2 | 0 | 2
  Abdomen | 1 | 0 | 1
  Appearance | 0 | 1 | 1
  Head, Eyes, Ears, Nose, Throat | 1 | 0 | 1
  Heart | 1 | 0 | 1
  Lungs | 1 | 0 | 1
  Vascular | 1 | 0 | 1
  Breasts | 0 | 0 | 0
  Chest | 0 | 0 | 0
  Lymph Nodes | 0 | 0 | 0
  Neurologic | 0 | 0 | 0
  Pelvis | 0 | 0 | 0
  Rectal | 0 | 0 | 0
  Thyroid | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: EGFR Phosphorylation in Normal Appearing Bladder Epithelium Adjacent to Tumor
Description: EGFR phosphorylation will be assessed using Immunohistochemistry (IHC), greater mean optical density is associated with greater phosphorylation. The difference between the placebo group and the erlotinib hydrochloride group will be tested as-randomized using a two-sample t-test with normalizing transformation if necessary or Wilcoxon rank-sum test.
Time Frame: Up to 18 hours after last study drug dose (on day 28)
Population: Number analyzed differs from number of participants in each arm for two reasons: sample size insufficient for analysis and sample not obtained.
Measure: Mean (Standard Deviation); unit: optical density
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Number analyzed (Participants) | 15 | 8
optical density
  Nucleus P-EGFR in Benign Tissue | 0.216 (0.063) | 0.181 (0.073)
  Cytoplasm P-EGFR in Benign Tissue | 0.159 (0.046) | 0.133 (0.062)
  Membrane P-EGFR in Benign Tissue | 0.179 (0.053) | 0.148 (0.074)
  Entire Cell P-EGFR in Benign Tissue | 0.190 (0.054) | 0.159 (0.069)
Statistical Analysis 1: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Nucleus P-EGFR in benign tissue between erlotinib and placebo; Test type: Other; p = 0.208, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Cytoplasm P-EGFR in benign tissue between erlotinib and placebo; Test type: Other; p = 0.208, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Membrane P-EGFR in benign tissue between erlotinib and placebo; Test type: Other; p = 0.272, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Entire Cell P-EGFR in benign tissue between erlotinib and placebo; Test type: Other; p = 0.220, Wilcoxon rank-sum test

2. Secondary Outcome: EGFR Phosphorylation in Neoplastic Bladder Epithelium 9-18 Hours Post-study Dose
Description: EGFR phosphorylation will be assessed using Immunohistochemistry (IHC), greater mean optical density is associated with greater phosphorylation.
Time Frame: Up to 18 hours after last study drug dose (on day 28)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Optical Density (OD)
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Number analyzed (Participants) | 21 | 11
Optical Density (OD)
  Nucleus P-EGFR Tumor Tissue | 0.175 (0.060) | 0.155 (0.059)
  Cytoplasm P-EGFR Tumor Tissue | 0.161 (0.053) | 0.146 (0.070)
  Membrane P-EGFR Tumor Tissue | 0.170 (0.058) | 0.154 (0.072)
  Entire Cell P-EGFR Tumor Tissue | 0.170 (0.056) | 0.151 (0.061)
Statistical Analysis 1: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Nucleus P-EGFR in Tumor Tissue, p-value between placebo and Erlotinib; Test type: Other; p = 0.361, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Cytoplasm P-EGFR in Tumor Tissue, p-value between placebo and Erlotinib; Test type: Other; p = 0.383, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Membrane P-EGFR in Tumor Tissue, p-value between placebo and Erlotinib; Test type: Other; p = 0.427, Wilcoxon rank-sum test
Statistical Analysis 4: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Entire Cell P-EGFR in Tumor Tissue, p-value between placebo and Erlotinib; Test type: Other; p = 0.416, Wilcoxon rank-sum test

3. Secondary Outcome: Pharmacokinetic Parameters: Erlotinib in Blood
Description: Will be summarized by treatment arm (and, if applicable, by visit) with appropriate descriptive statistics.
Time Frame: Baseline, day 8, and day 16 (day of surgery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Number analyzed (Participants) | 24 | 13
ng/mL
  Baseline | 0.0 (0.0) | 0.0 (0.0)
  Day 8: number analyzed (Participants) | 13 | 5
  Day 8 | 169.7 (581.3) | 0.0 (0.0)
  Day 16 (Surgery): number analyzed (Participants) | 24 | 11
  Day 16 (Surgery) | 2218.4 (1096.1) | 0.3 (1.2)
Statistical Analysis 1: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Baseline visit - p-value between erlotinib and placebo arms; Test type: Other; p = 1.000, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Day 8 - p-value between erlotinib and placebo arms; Test type: Other; p = 0.199, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Surgery visit - p-value between erlotinib and placebo arms; Test type: Other; p < 0.001, Wilcoxon rank-sum test

4. Secondary Outcome: Pharmacokinetic Parameters: OSI-420 in Blood
Description: Will be summarized by treatment arm (and, if applicable, by visit) with appropriate descriptive statistics.
Time Frame: Baseline, day 8, and day 16 (day of surgery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Number analyzed (Participants) | 24 | 13
ng/mL
  Baseline | 0.0 (0.0) | 0.0 (0.0)
  Day 8: number analyzed (Participants) | 13 | 5
  Day 8 | 2.5 (7.3) | 0.0 (0.0)
  Day 16 (Surgery): number analyzed (Participants) | 24 | 11
  Day 16 (Surgery) | 44.4 (34.6) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Baseline visit - p-value between erlotinib and placebo arms; Test type: Other; p = 1.000, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Day 8 - p-value between erlotinib and placebo arms; Test type: Other; p = 0.288, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Surgery visit - p-value between erlotinib and placebo arms; Test type: Other; p < 0.001, Wilcoxon rank-sum test

5. Secondary Outcome: Frequency of Urination Symptoms in Men Only, Graded According to International Prostate Symptom Score (I-PSS)
Description: A well documented survey called the International Prostate Symptom Score (I-PSS) of urination symptoms which correlates with prostatic hyperplasia in men will be filled out by men at baseline and end of study. The I-PSS is an 8-item survey; 7 questions scored from 0-5 where 0 is 'none' or 'not at all' and 5 is 'five times' or 'almost always'. The sum of the scores for the first 7 questions has a total range of 0-35 where 0 is asymptomatic, 1-7 is mild symptoms, 8-19 is moderate symptoms, and 20-35 are severe symptoms. A final quality of life question is scored from 0-6 where 0 (delighted) to 6 (terrible). This question serves as a conversation starting point between the patient and physician.
Time Frame: Baseline up to 18 hours after last study drug dose (on day 28)
Population: A participant in the placebo group had no survey response at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Number analyzed (Participants) | 15 | 7
Participants
  Baseline: number analyzed (Participants) | 15 | 6
  Baseline: Mild (score of 1-7) | 7 | 3
  Baseline: Moderate (score of 8-19) | 7 | 3
  Baseline: Severe (score of 20-35) | 1 | 0
  Surgery Visit: Mild (score of 1-7) | 7 | 5
  Surgery Visit: Moderate (score of 8-19) | 7 | 2
  Surgery Visit: Severe (score of 20-35) | 1 | 0
Statistical Analysis 1: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); P-value between groups at Baseline; Test type: Other; p = 0.792, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); P-value between groups at surgery visit; Test type: Other; p = 0.261, Wilcoxon rank-sum test

6. Secondary Outcome: Expression of E-cadherin
Description: E-Cadherin expression will be assessed using Immunohistochemistry (IHC), greater membrane optical density was associated with greater expression. A two-sample t-test with normalizing transformation if necessary or Wilcoxon rank-sum test will be used.
Time Frame: At time of surgery (approximately day 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Optical Density (OD)
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Number analyzed (Participants) | 15 | 9
Optical Density (OD)
  Benign Tissue | 0.615 (0.126) | 0.572 (0.198)
  Tumor Tissue | 0.616 (0.070) | 0.563 (0.079)
Statistical Analysis 1: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Expression of e-cadherin in Benign Tissue, P-Value between arms; Test type: Other; p = 0.721, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Expression of e-cadherin in Tumor Tissue, P-Value between arms; Test type: Other; p = 0.108, Wilcoxon rank-sum test

7. Secondary Outcome: Percentage of Cells Expressing Ki67
Description: Ki-67 expression will be assessed using Immunohistochemistry (IHC), greater positivity was associated with greater expression. A two-sample t-test with normalizing transformation if necessary or Wilcoxon rank-sum test will be used.
Time Frame: At time of surgery (approximately day 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Number analyzed (Participants) | 15 | 9
percentage
  Benign Tissue | 0.093 (0.142) | 0.080 (0.111)
  Tumor Tissue | 0.148 (0.142) | 0.170 (0.137)
Statistical Analysis 1: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Expression of KI-67 in Benign Tissue, P-Value between arms; Test type: Other; p = 0.444, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Expression of KI-67 in Tumor Tissue, P-Value between arms; Test type: Other; p = 0.663, Wilcoxon rank-sum test

8. Secondary Outcome: Difference Between Normal and Neoplastic Tissue Phosphorylated ERK
Description: Phosphorylated ERK will be assessed using Immunohistochemistry (IHC), greater mean optical density is associated with greater expression. A two-sample t-test with normalizing transformation if necessary or Wilcoxon rank-sum test will be used.
Time Frame: At time of surgery (approximately day 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Optical Density (OD)
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Number analyzed (Participants) | 12 | 5
Optical Density (OD)
  Nucleus P-ERK Normal-Tumor | -0.071 (0.167) | -0.077 (0.183)
  Cytoplasm P-ERK Normal-Tumor | -0.104 (0.187) | -0.098 (0.170)
  Entire Cell P-ERK Normal-Tumor | -0.084 (0.171) | -0.085 (0.173)
Statistical Analysis 1: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Difference in p-ERK between Normal and Tumor Tissue, P-Value between arms; Test type: Other; p = 1.000, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Difference in Cytoplasm p-ERK between Normal and Tumor Tissue, P-Value between arms; Test type: Other; p = 0.792, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Difference in Entire Cell p-ERK between Normal and Tumor Tissue, p-value between arms; Test type: Other; p = 1.000, Wilcoxon rank-sum test

9. Secondary Outcome: Difference Between Normal and Neoplastic Tissue of p53
Description: p53 expression will be assessed using Immunohistochemistry (IHC), greater nucleus optical density and positivity was associated with greater expression. A two-sample t-test with normalizing transformation if necessary or Wilcoxon rank-sum test will be used.
Time Frame: At time of surgery (approximately day 16)
Population: Number analyzed differs from number of participants in each arm for two reasons: sample size insufficient for analysis and sample not obtained. As well as there was not enough tissue to complete this analysis for all participants.
Measure: Mean (Standard Deviation); unit: Optical Density (OD)
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Number analyzed (Participants) | 13 | 8
Optical Density (OD) | -0.052 (0.185) | -0.115 (0.305)
Statistical Analysis 1: Comparison: Group I (Erlotinib Hydrochloride) vs Group II (Placebo); Test type: Other; p = 0.772, Wilcoxon rank-sum test

10. Secondary Outcome: Difference Between Normal and Neoplastic Tissue of Let-7
Description: A two-sample t-test with normalizing transformation if necessary or Wilcoxon rank-sum test will be used.
Time Frame: At time of surgery (approximately day 16)
Population: This analysis was not completed after discussions with DCP. Participant samples were rationed for multiple analyses, Let-7 analysis was determined to be low on the priority list and it was decided to forego this analysis.
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 9 weeks
Arm/Group | Group I (Erlotinib Hydrochloride) | Group II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/24 | 2/13
Other Adverse Events (participants affected / at risk) | 22/24 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Erlotinib Hydrochloride) (N=24) | Group II (Placebo) (N=13)
Surgical and Medical Procedures, Other (Surgical and medical procedures) | 0 (0) | 2 (2)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Erlotinib Hydrochloride) (N=24) | Group II (Placebo) (N=13)
Blood and Lymphatic System Disorders, Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymph Node Pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Endocrine Orders, Other (Endocrine disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 9 (13) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal Disorders, Other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2)
Infections and Infestations, Other (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 2 (2) | 0 (0)
Investigations, Other (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and Connective Tissues Disorder, Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive Disturbance (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Bladder Spasm (Renal and urinary disorders) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary Tract Pain (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary Urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, Thoracic, and Mediastinal Disorders, Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 6 (11) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Scalp Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and Subcuteaneous Tissue Disorders, Other (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Surgical and Medical Procedures, Other (Surgical and medical procedures) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hot Flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 9 (11) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT02169284/Prot_SAP_000.pdf